CLINICAL TRIAL: NCT04137133
Title: Patienthèque of Finisterian (South of Brittany) Children With Cystic Fibrosis in the Time of Precision Medicine.Descriptive Monocentric Study for Identification and Validation of Biomarkers Predictive of Clinical Evolution
Brief Title: Patienthèque of Finisterian (South of Brittany) Children With Cystic Fibrosis in the Time of Precision Medicine
Acronym: MUCOthèque
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MUCOthèque (29BRC19.0102)
Record Dates: First submitted 2019-10-22; First posted 2019-10-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- collection of expectoration, stools and blood (Experimental)
  Interventions: Diagnostic Test: collection

INTERVENTIONS:
Diagnostic Test: collection — bronchial secretions, blood, stools, superficial skin sample, dental plaque sample and urine

SUMMARY:
The objective of this study is to evaluate the relevance of Porphyromonas as a biomarker predicting the risk of P. aeruginosa primocolonization in children form 0 to 18 years old with cystic fibrosis.

DETAILED DESCRIPTION:
This is a monocentric study in 3 phases:

* Pre-inclusion: at the first visit to the CRCM (support for a positive screening confirmed by sweat test and genotyping CFTR)
* Inclusion: possible between the 2nd visit to the CRCM (about 2 months old) and the 6th month
* Follow-up: up to 36 months old. The pace of visits will be based on the usual follow-up rate of CF infants Clinical and paraclinical data and samples will be collected as part of the usual follow-up of CF children. Inclusions and follow-up visits will be carried out at the Roscoff CRCM as well as respiratory explorations and biological samples. Dermatological and odontological follow-ups will be scheduled for each patient at the rate of an annual visit to the CHRU in Brest in the relevant departments.

ELIGIBILITY:
Inclusion Criteria:

* Newly screened infants with a confirmed diagnosis of cystic fibrosis in its classic form (clinical symptoms and two positive sweat tests and/or two mutations of the cftr gene from Class I to III)
* Children free of any colonization with P. aeruginosa
* Affiliation with the social security system
* Consent signed by the holders of parental authority or the sole parent holding parental authority

Exclusion Criteria:

* Children colonized with P. aeruginosa according to the cytobacteriological examination and / or molecular test of sputum or pharyngeal specimens
* Children grafted
* Children not affiliated to a social security scheme or not entitled to
* Children whose parent (s) are (are) minor (s)
* Children whose holders of parental authority do not master the French language
* Refusal to participate in the study

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-03-21 (Actual); Primary Completion 2030-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Presence of P. aeruginosa in bacterial sputum cultures in one of bronchial secretions sample | 3 years
  Analyse with Porphyromonas predictive biomarker of the risk of P. aeruginosa primocolonization.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ildys, Roscoff, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending fifteen years following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.